CLINICAL TRIAL: NCT05430620
Title: A Prospective Feasibility Trail to Compare the Efficacy of Intermittent Surface Oxygenation With Continuous Surface Oxygenation During Hypothermic Machine Perfusion of Kidneys Donated After Circulatory Death
Brief Title: Intermittent Versus Continuous Surface O2 During HMP of DCD Kidneys
Acronym: HMPO2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/21MAI/239
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Delayed Graft Function; Kidney Transplant; Complications; Ischemia Reperfusion Injury; Mitochondrial
Keywords: Hypothermic oxygenated machine perfusion; Kidney preservation; bubble and surface oxygenation
MeSH Terms: conditions — Delayed Graft Function; Reperfusion Injury | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Kidneys originating from deceased donors after circulatory death (DCD), category 3 and 5 (controlled) will be preserved from procurement until transplantation on hypothermic machine perfusion conditions and prospectively randomized into 2 study groups: 1) intermittent surface oxygenation during HMP (surface oxygenation interrupted during organ transport (2-4h)(I-HMPO2 group), and 2) continuous surface oxygenation during HMP (surface oxygenation during the whole machine preservation period included organ transport)(C-HMPO2 group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I-HMPO2 (Experimental): intermittent surface oxygenation during hypothermic machine perfusion (surface oxygenation interrupted during organ transport)
  Interventions: Drug: Oxygen
- C-HMPO2 (Active Comparator): continuous surface oxygenation during HMP (surface oxygenation during the whole machine preservation period included organ transport)
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Active oxygenation during hypothermic machine perfusion by bubble and surface oxygenation. Intermittent surface oxygenation is compared with continuous surface oxygenation during hypothermic machine perfusion
  Other Names: feasibility of bubble and surface oxygenation applied to the LifePort Kidney Transporter (Organ Recovery Systems, Diegem, Belgium)

SUMMARY:
The aim of the study is to evaluate the feasibility of this bubble and surface oxygenation and to determine the optimal timing of surface oxygenation (continuous versus intermittent) as alternative for membrane-oxygenated kidneys, originating from DCD donors, during HMP on early graft function in clinical practice.

DETAILED DESCRIPTION:
Kidneys originating from deceased donors after circulatory death (DCD), category 3 and 5 (controlled) will be preserved from procurement until transplantation on hypothermic machine perfusion conditions and prospectively randomized into 2 study groups: 1) intermittent surface oxygenation during HMP (surface oxygenation interrupted during organ transport (2-4h)(I-HMPO2 group), and 2) continuous surface oxygenation during HMP (surface oxygenation during the whole machine preservation period included organ transport)(C-HMPO2 group).

ELIGIBILITY:
Inclusion Criteria:

* Listed for a renal transplantation due to end stage renal disease
* Willingness to comply with the protocol procedures for the duration of the study included scheduled follow-up visits and examinations.

Exclusion Criteria:

* Multi-organ recipients
* Dual kidney transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Functional delayed graft function | first 7 days after transplantation
  defined as the absence of a decrease in the serum creatinine level of at least 10% per day for at least 3 consecutive days in the first 7 days after transplantation (not including patients in whom acute rejection of calcineurin inhibitor toxicity is proven on biopsy)

SECONDARY OUTCOMES:
Need for dialysis after transplantation | 0-30 days after transplantation
  Number of dialysis sessions after transplantation
Delayed graft function | first 7 days after transplantation
  defined as the need for dialysis in the first 7 days after transplantation and preceding the return of kidney function
Serum creatinine reduction ratio | Day 1-2 after transplantation
  alternative definition of DGF= CRR2 < or = 30%
Graft survival | From 1-365 days after transplantation
  Functional kidney graft at 7 days, 3, 6, and 12 months
Patient survival (censored and uncensored for death) | From 1-365 days after transplantation
  Patient survival at 7 days, 3, 6, and 12 months
Glomerular filtration rate at 1 year after transplantation | At 1 year after transplantation (window 30 days)
  24-hour creatinine clearance
Estimated glomerular filtration rate | At 3, 6, and 12 months after transplantation with window of 10 days
  eGFR defined by the CKD-EPI equation (Chronic Kidney Disease Epidemiology Collaboration) at 3, 6 and 12 months after transplantation
Primary non-function | Until 3 months after transplantation
  defined as the continued need for dialysis at 3 months after transplantation
Biopsy-proven acute rejection | Until 1 year after transplantation with window of 10 days
  Biopsy-proven acute rejection during the 1 year after transplantation
Metabolic analysis on kidney preservation tissue | Baseline and pre-surgery
  Metabolic analysis by 1D proton NMR (e.g., succinate, lactate, acetate, formate, hypoxanthine) on a tissue sample taken before (= baseline) and at the end of the preservation period before transplantation of the kidney
Metabolic analysis on kidney preservation tissue | Baseline and pre-surgery
  Metabolic analysis by liquid chromatography coupled to electrospray ionization mass spectrometry (LC-ESI-MS) (succinate, glutamate, lactate, ATP, ADP, AMP, NADH, NAD+) on a tissue sample taken before (= baseline) and at the end of the preservation period before transplantation of the kidney
Metabolic analysis on preservation fluid | Baseline and pre-surgery
  Metabolic analysis by 1D proton NMR and fluorescence on a perfusion fluid sample taken before (= baseline) and at the end of the preservation period before transplantation of the kidney

CONTACTS AND LOCATIONS:
Overall Officials: Tom Darius, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Woluwé-Saint-Lambert, Belgium

IPD SHARING:
Plan to Share IPD: No